CLINICAL TRIAL: NCT04384692
Title: Peritransplant Ruxolitinib for Patients With Primary and Secondary Myelofibrosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1006507; NCI-2020-01626 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10093 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Primary Myelofibrosis; Secondary Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — Stem Cell Transplantation; Busulfan; Cyclophosphamide; fludarabine; Melphalan; Methotrexate; merphos; Mycophenolic Acid; ruxolitinib; Tacrolimus; Whole-Body Irradiation; Biopsy; Magnetic Resonance Spectroscopy; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ruxolitinib, conditioning, HSCT, GVHD prophylaxis) (Experimental): See detailed description.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Busulfan; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Melphalan; Drug: Methotrexate; Drug: Mycophenolate Mofetil; Drug: Ruxolitinib; Drug: Tacrolimus; Radiation: Total-Body Irradiation; Procedure: Computed Tomography; Procedure: Echocardiography; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo HSCT
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039; Jylamvo
Drug: Mycophenolate Mofetil — Given IV or PO
  Other Names: CellCept; MMF
Drug: Ruxolitinib — Given PO
  Other Names: INCB-18424; INCB18424; Oral JAK Inhibitor INCB18424
Drug: Tacrolimus — Given IV and PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TBI; Total Body Irradiation; Whole Body Irradiation; Whole-Body Irradiation; Total-Body Irradiation Prior to Stem Cell Transplant
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT Scan; Computed Axial Tomography
Procedure: Echocardiography — Undergo echocardiography
  Other Names: EC
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration and biopsy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MRI
Procedure: Ultrasound Imaging — Undergo ultrasound imaging
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging

SUMMARY:
This phase II trial studies how well administering ruxolitinib before, during, and after allogeneic hematopoietic stem cell transplantation works in preventing graft versus host disease and improving transplant outcomes in patients with primary and secondary myelofibrosis. Donor hematopoietic stem cell transplantation (HSCT) is currently the only treatment with proven curative potential for myelofibrosis, however, myelofibrosis patients have a high risk for developing graft versus host disease post-transplant. Graft versus host disease is a condition where the transplanted cells from a donor can attack the body's normal cells. Ruxolitinib, a janus-associated kinase (JAK) inhibitor, is known to decrease inflammatory signals, which may reduce spleen size and decrease symptoms such as night sweats and weight loss. Administering ruxolitinib before, during, and after transplant may decrease the incidence and severity of graft versus host disease, increase survival, and improve quality of life in patients with primary and secondary myelofibrosis.

DETAILED DESCRIPTION:
OUTLINE:

PART 1: Patients receive ruxolitinib orally (PO) starting 8 weeks prior to hematopoietic stem cell transplantation (HSCT) and continuing until approximately 14 days prior to conditioning regimen, then tapered per the treating clinician until day -4 in the absence of disease progression or unacceptable toxicity. Patients who join a different research study for Part 2 have their collected data and samples from Part 1 carried over to the new protocol.

PART 2: Patients are assigned to either a high (myeloablative) or reduced intensity conditioning regimens per the clinical provider together with the Clinical Coordinators Office (CCO):

MYELOABLATIVE CONDITIONING: Patients receive cyclophosphamide intravenously (IV) on days -7 and -6 and busulfan IV over 3 hours on days -5 to -2. Patients with umbilical cord blood (UCB) as their transplant source also receive fludarabine IV over 30 minutes on days -8 to -6. Treatment continues in the absence of disease progression or unacceptable toxicity.

REDUCED INTENSITY CONDITIONING: Patients receive fludarabine IV over 30 minutes on days -6 to -2 and melphalan IV over 15-30 minutes on days -3 and -2. Patients with UCB as their transplant source also undergo total body irradiation (TBI) on day -1. Treatment continues in the absence of disease progression or unacceptable toxicity.

TRANSPLANT: After completion of conditioning regimen, patients undergo HSCT on day 0.

GVHD PROPHYLAXIS: Patients receive ruxolitinib until approximately 7 months post-transplant and then tapered over 2 months until 9-12 months post HSCT. Patients also receive tacrolimus IV continuously (inpatients) or every 12 hours (outpatients) beginning day -1 (day -3 for patients with UCB as their donor source), then PO twice daily (BID) once therapeutic levels are reached, with a taper beginning on day 56 for patients with related donors, and day 100 for patients with unrelated donors over 4 months in the absence of GVHD. The duration of tacrolimus for patients with GVHD is determined by the attending physician. Patients with related and unrelated donors also receive methotrexate IV on days 1, 3, 6, and 11. Patients with UCB as their transplant source also receive mycophenolate mofetil IV or PO every 8 hours beginning on days 0-30, then tapered until day 40 in the absence of GVHD. All treatment continues in the absence of disease progression or unacceptable toxicity.

Patients undergo computed tomography (CT) scan and may undergo echocardiography on study and bone marrow aspiration and biopsy and blood sample collection and may undergo magneti resonance imaging (MRI) and ultrasound throughout the study.

Patients are followed up at 6 months, 1 year, and 2-5 years after completion of HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* JAK INHIBITOR ADMINISTRATION INCLUSION: (PART I)
* Disease criteria:

  * Diagnosis of primary myelofibrosis (PMF) as defined by the 2016 World Health Organization classification system or diagnosis of secondary myelofibrosis (MF) as defined by the International Working Group (IWG) for Myeloproliferative Neoplasms Research and Treatment criteria
  * Patients meeting the criteria for intermediate-1, intermediate-2 or high-risk disease by Dynamic International Prognostic Scoring System (DIPSS) or DIPSS plus
* Ability to understand and the willingness to sign a written informed consent document
* Patient must be a potential hematopoietic stem cell transplant candidate as assessed by the consenting physician
* Patient must be willing to start ruxolitinib within a 6-month time period
* ALLOGENEIC STEM CELL TRANSPLANT INCLUSION: (PART II)
* Meeting criteria for part 1, as above, at time of initiation of ruxolitinib, including the ability to understand and willingness to sign a written informed consent. Patients arriving to our institution for transplant and not enrolled in part 1 may still be enrolled in part 2 if part 1 criteria are met. These patients will have part 1 endpoints transcribed from medical records
* Received ruxolitinib for at least 8 weeks immediately prior to conditioning and be willing to continue until 9-12 months post-transplant as tolerated
* Performance status score: Karnofsky >= 70
* Calculated creatinine clearance using the Cockcroft-Gault formula or 24 hour (hr) urine creatinine clearance must be > 60 ml/min
* Total serum bilirubin must be < 3 mg/dL unless the elevation is thought to be due to Gilbert's disease or hemolysis
* Transaminases must be < 3 x the upper limit of normal
* Patients with clinical or laboratory evidence of liver disease will be evaluated for the cause of liver disease, its clinical severity in terms of liver function, and the degree of portal hypertension. Patients with fulminant liver failure, cirrhosis with evidence of portal hypertension or bridging fibrosis, alcoholic hepatitis, hepatic encephalopathy, or correctable hepatic synthetic dysfunction evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3mg/dL, and symptomatic biliary disease will be excluded
* Diffusion capacity of lung for carbon monoxide (DLCO) corrected > 60% normal. May be not be on supplemental oxygen
* Left ventricular ejection fraction > 40% OR shortening fraction > 26%
* Comorbidity index < 5 at the time of pre-transplant evaluation

Exclusion Criteria:

* JAK INHIBITOR ADMINISTRATION EXCLUSION: (PART I)
* Contraindication to receiving ruxolitinib including:

  * Patients who have known hypersensitivity to JAK inhibitors
  * Clinical or laboratory evidence of significant renal or hepatic impairment including cirrhosis
  * Active uncontrolled infection
  * Known human immunodeficiency virus (HIV) positivity
  * Women who are pregnant or trying to conceive
  * Caution should be used in patients with platelets < 100 though adjustments in dose can be made to accommodate anyone with platelets > 50
* History of prior allogeneic transplant
* Leukemic transformation (> 20% blasts)
* ALLOGENEIC STEM CELL TRANSPLANT EXCLUSION: (PART II)
* Uncontrolled viral or bacterial infection at the time of transplant data review and consent conference
* Active or recent (prior 6 month) invasive fungal infection without infectious disease (ID) consult and approval
* History of HIV infection
* Pregnant or breastfeeding
* Patients without a human leukocyte antigen (HLA)-identical sibling donor, 10 of 10 HLA-matched or 9 of 10 allele mismatched unrelated donor, or umbilical cord blood units that meet transplant criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2030-04-23 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade II-IV graft versus host disease (GVHD) in myelofibrosis patients | Up to day 100
  The probability of grade II-IV acute GVHD observed in this study will be compared to a fixed benchmark, this fixed benchmark derived from the results of a previous study (FH Protocol 9033).

SECONDARY OUTCOMES:
Incidence of grade III-IV GVHD | Up to day 100
  Estimated as simple proportions and informally compared to the results from FH Protocol 9033.
Incidence of chronic GVHD | At 1 and 2 years
Overall survival rate (OS) | At 1 and 2 years
Incidence of primary and secondary graft failure | 6 months
  Estimated as simple proportions and informally compared to the results from FH Protocol 9033.
Time to neutrophil (ANC > 500) engraftment | Day 100
Time to platelet (> 20,000) engraftment | Day 100
Incidence of relapse | At 1 year
Non-relapse mortality (NRM) | Day 100 and 1 year
  Estimated as simple proportions and informally compared to the results from FH Protocol 9033.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel B. Salit, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-02-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT04384692/ICF_000.pdf